CLINICAL TRIAL: NCT06863688
Title: Does Tourniquet Utilization Negatively Impact Patient Pain and Outcomes Following Operative Fixation of Rotational Ankle Fractures? a Randomized Clinical Trial.
Brief Title: Ankle Fracture Tourniquet Utilization
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Alex Demers (Other)
Responsible Party: Sponsor-Investigator, Alex Demers, Resident Physician, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202311372
Record Dates: First submitted 2025-01-05; First posted 2025-03-07 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-01

CONDITIONS: Ankle Fracture
Keywords: Ankle Fracture; Tourniquet; PROM; Pain
MeSH Terms: conditions — Ankle Fractures; Pain | interventions — Tourniquets

STUDY DESIGN:
Intervention Model Description: Patients undergoing operative fixation of ankle fractures will be randomized to the tourniquet and no tourniquet groups in a 1:1 fashion. The treating orthopaedic trauma surgeon will be informed of the randomization status the day of surgery by the PI to ensure appropriate tourniquet utilization is executed during surgery.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tourniquet Group (Experimental): Patients randomized to this group will have a tourniquet used during the operative fixation of their ankle fracture. Tourniquets will be inflated to 250 mmHg as is standard for our institution. Tourniquet will be deflated at time of closure.
  Interventions: Device: Tourniquet
- No Tourniquet Group (Other): Patients randomized to this group will not have a tourniquet used during operative fixation of their ankle fracture. A tourniquet will be placed on the patient's operative extremity as a safety precaution, but will remain deflated for the duration of the procedure unless emergently needed for hemostasis.
  Interventions: Other: No Tourniquet

INTERVENTIONS:
Device: Tourniquet — Tourniquets will be applied to the thigh of the operative extremity during operative fixation of ankle fractures.
  Arms: Tourniquet Group
Other: No Tourniquet — No tourniquet will be inflated on the operative extremity during the operative fixation of ankle fractures.
  Arms: No Tourniquet Group

SUMMARY:
Lower extremity tourniquet utilization remains a controversial practice during the operative fixation of rotational ankle fractures and is often left to surgeon discretion. At our own institution, tourniquet use varies between surgeons with some providers using a tourniquet for every case, while others regularly do not utilize tourniquets. Despite benefits of decreased surgical time and decreased blood loss, many studies have cited negative outcomes associated with tourniquet usage including increased postoperative swelling and pain, increased wound complications, and increased risks of deep vein thrombosis. These outcomes have been limited to retrospective reviews and meta-analyses with few randomized control trials specifically evaluating these outcomes in ankle fracture patients. To better assess the impact of tourniquet use on ankle fracture postoperative outcomes, this randomized control trial seeks to 1) compare differences in postoperative visual analog scale pain scores for patients undergoing operative fixation of rotation ankle fractures with and without a tourniquet, while 2) evaluating rates of wound, thrombotic, and surgical complications associated with tourniquet use. Patients will be randomized by an Excel random number generator to a tourniquet and non-tourniquet group. Patients will remain blinded to randomization. The treating orthopaedic trauma surgeon will be notified by the PI of the study informing them of the randomization status to ensure appropriate tourniquet utilization the day of surgery. Patients will then undergo standard operative fixation and postoperative management as clinically indicated by the orthopaedic trauma team. Patients will follow-up at 2 weeks and subsequently every 4 weeks as is protocol at our institution. Patient charts will be reviewed for patient and perioperative factors, as well as postoperative complications (i.e. wound complications, need for repeat surgical intervention, and deep vein thrombosis).

DETAILED DESCRIPTION:
Lower extremity tourniquet utilization remains a controversial practice during the operative fixation of rotational ankle fractures and is often left to surgeon discretion. At our own institution, tourniquet use varies between surgeons with some providers using a tourniquet for every case, while others regularly do not utilize tourniquets. Despite benefits of decreased surgical time and decreased blood loss, many studies have cited negative outcomes associated with tourniquet usage including increased postoperative swelling and pain, increased wound complications, and increased risks of deep vein thrombosis. These outcomes have been limited to retrospective reviews and meta-analyses with few randomized control trials specifically evaluating these outcomes in ankle fracture patients. To better assess the impact of tourniquet use on ankle fracture postoperative outcomes, this randomized control trial seeks to 1) compare differences in postoperative visual analog scale pain scores for patients undergoing operative fixation of rotation ankle fractures with and without a tourniquet, while 2) evaluating rates of wound, thrombotic, and surgical complications associated with tourniquet use. II.

Tourniquet utilization in the operative fixation of ankle fractures remains controversial and is often subject to surgeon preferences. Despite postulated benefits of minimizing blood loss, decreasing operative times, and improving visualization, tourniquets in ankle fracture fixation have been associated with increased postoperative pain, swelling, decreased range of motion, and increased opioid consumption. Previous literature has demonstrated a nonsignificant increase in wound infections and deep vein thrombosis (DVT) with tourniquet usage. Changes in perfusion intraoperatively and effects of ischemic reperfusion injury have been theorized as drivers of these negative side effects of tourniquets. Perfusion following ankle fracture fixation, thus represents an opportunity to better understand the physiologic implications of tourniquet utilization.

Tourniquet use is associated with negative outcomes after total knee arthroplasty (TKA). Despite decreased blood loss, tourniquet use in TKA has been associated with higher VAS pain scores, decreased knee range of motion and functional scores in the early postoperative period, higher rates of thrombotic events, infection, and reoperation. Impaired prosthesis survival, knee function, blood transfusion rates, quality of life, and patient satisfaction bring into question the utility of tourniquet use in TKA. These outcomes have not been thoroughly investigated in the fixation of ankle fractures.

ELIGIBILITY:
Inclusion criteria:

1. Patients >18 y.o. undergoing ankle fracture open reduction internal fixation
2. Ground level fall as mechanism of injury
3. Closed injury

Exclusion criteria:

1. Open Ankle Fractures
2. Vascular Injury Requiring Intervention
3. Lower extremity injuries on same side of ankle fracture

e) Active anticoagulation/bleeding disorder necessitating tourniquet use (Hemoglobin <7, PT >13, PTT>35) f) Ipsilateral lower extremity trauma impacting immobilization g) Patients with peripheral neuropathy h) Patients undergoing ankle arthroscopy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale Pain Levels | Post anesthesia recovery unit, 2 weeks postoperatively, 3 month follow-up
  VAS pain scores (0-10) will be assessed for the ankle immediately postoperatively in the post anesthesia care unit and at 2 weeks and 3 months postoperatively.
Patient-Reported Outcome Measurement Information System (PROMIS) Cat V1.1 Pain Interference scores | 6 weeks, 3 months
  Patient-Reported Outcome Measurement Information System (PROMIS) scores including PROMIS Cat V1.1 Pain Interference (10-90, lower is better) will be completed at 6 week and 3 month follow-up appointments as part of standard clinic workflow.
Patient-Reported Outcome Measurement Information System (PROMIS) Cat V2.0 Physical Function Score | 6 weeks, 3 month
  Patient-Reported Outcome Measurement Information System (PROMIS) scores including PROMIS Cat V2.0 Physical Function (10-90, higher is better) will be completed at 6 week and 3 month follow-up appointments as part of standard clinic workflow.
Patient-Reported Outcome Measurement Information System (PROMIS) Scale V1.2 Global Health Score | 6 weeks, 3 months
  Patient-Reported Outcome Measurement Information System (PROMIS) scores including PROMIS Scale V1.2 Global Health (15-70, higher is better) will be completed at 6 week and 3 month follow-up appointments as part of standard clinic workflow.
Optimal Screening for Prediction of Referral and Outcome (OSPRO) Yellow Flag 17-Item | 2 weeks, 6 weeks, 3 months
  OSPRO-Yf 17 questionnaires will be completed at follow-up appointments as part of standard trauma clinic workflow and will be assessed at 2 weeks, 6 weeks, and 3 months.

SECONDARY OUTCOMES:
Postoperative Complications | 6 months
  Postoperative complications following operative fixation of ankle fractures will be assessed at follow-up appointments and through chart review. Complications include postoperative deep vein thrombosis, wound complications and infection (patients receiving antibiotics or requiring surgical irrigation and debridement), need for revision fixation or hardware removal.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Demers, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared secondary to data sharing regulations at our institution.

REFERENCES:
- [Background] Zhang W, Li N, Chen S, Tan Y, Al-Aidaros M, Chen L. The effects of a tourniquet used in total knee arthroplasty: a meta-analysis. J Orthop Surg Res. 2014 Mar 6;9(1):13. doi: 10.1186/1749-799X-9-13. PMID 24602486
- [Background] Benedick A, Rivera T, Vallier HA. Effect of Tourniquet Use During Ankle Fracture Fixation on Wound Healing and Infectious Complications. Foot Ankle Int. 2020 Jun;41(6):714-720. doi: 10.1177/1071100720907379. Epub 2020 Mar 1. PMID 32116012
- [Background] Konrad G, Markmiller M, Lenich A, Mayr E, Ruter A. Tourniquets may increase postoperative swelling and pain after internal fixation of ankle fractures. Clin Orthop Relat Res. 2005 Apr;(433):189-94. doi: 10.1097/01.blo.0000151849.37260.0a. PMID 15805957
- [Background] Davey MS, Davey MG, Hurley ET, Kearns SR. Tourniquet Use During Open Reduction and Internal Fixation of Ankle Fractures - A Systematic Review and Meta-Analysis. J Foot Ankle Surg. 2022 Sep-Oct;61(5):1103-1108. doi: 10.1053/j.jfas.2022.01.019. Epub 2022 Jan 23. PMID 35219596
- [Background] Kruse H, Christensen KP, Moller AM, Gogenur I. Tourniquet use during ankle surgery leads to increased postoperative opioid use. J Clin Anesth. 2015 Aug;27(5):380-4. doi: 10.1016/j.jclinane.2015.03.034. Epub 2015 May 12. PMID 25979462
- [Background] Younger AS, Kalla TP, McEwen JA, Inkpen K. Survey of tourniquet use in orthopaedic foot and ankle surgery. Foot Ankle Int. 2005 Mar;26(3):208-17. doi: 10.1177/107110070502600305. PMID 15766423